CLINICAL TRIAL: NCT01844141
Title: Effectiveness of the Lavage With 70% Alcohol Plus 0.5% Chlorhexidine Compared to 70% Alcohol for Chemical Matricectomy in the Surgical Treatment of Ingrown Toenails
Brief Title: Effectiveness of Lavage With Alcohol - Chlorhexidine for Chemical Matricectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Ricardo Becerro de Bengoa Vallejo, PhD, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIC11022013
Record Dates: First submitted 2013-02-11; First posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Ingrown Toenail
Keywords: phenol; ingrown toenail; chemical matricectomy
MeSH Terms: conditions — Nails, Ingrown | interventions — Ethanol; Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alcohol - clorhexidine (Experimental): Ingrown toenail irrigated using 70% alcohol - 0.5% clorhexidine
  Interventions: Drug: 70% alcohol - 0.5% clorhexidine
- 70% alcohol (Active Comparator): Ingrown toenail irrigated using 70% alcohol
  Interventions: Drug: 70% alcohol

INTERVENTIONS:
Drug: 70% alcohol — After phenolization of the ingrown toenail the wound is irrigated with 15 cc solution of 70% alcohol plus 0.5% clorhexidine
  Other Names: Isopropilic alcohol.; Ethanol
  Arms: 70% alcohol
Drug: 70% alcohol - 0.5% clorhexidine — In the intervention group five rounds of 3 ml wash of 70% alcohol - 0.5% clorhexidine was used to irrigate the exposed area of the nail to neutralize any residual effect of phenol and found out how much residual phenol is still in the wound.
  Other Names: chlorhexidine-gluconate
  Arms: alcohol - clorhexidine

SUMMARY:
To compare the efficacy of the lavage with 70% alcohol plus 0.5% chlorhexidine versus 70% alcohol in the surgical treatment of ingrown toenails.

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy of the lavage with 70% alcohol plus 0.5% chlorhexidine versus 70% alcohol during the phenolization procedure in the surgical treatment of ingrown toenails in patients undergoing for chemical matricectomy.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 with onychocryptosis

Exclusion Criteria:

* infection, history of tinea pedis, onychomycosis, paronychia, nail trauma or subungual hematoma, nail deformities and disorders, peripheral vascular disease or diabetes, cardiac disease, history of rheumatic fever, recent antibiotic use or current antimicrobial therapy, history of steroid use and recent nail polish use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Quantity of phenol recovered in each lavage with each solution | up to 2 weeks
  The amounts of phenol in the samples were quantified by a Jasco modular high performance liquid chromatograph HPLC (Jasco International Co Ltd, Japan) equipped with a LG-2080-04 quaternary low-gradient unit, a PU-2080 pump, a DG-2080-54 degasser, an AS-2050-plus autosampler and a UV-2070 plus UV/Vis detector was used. A C18 column Luna (particle size 3 µm, 150 x 4.6 mm) (Phenomenex, Torrance, CA, USA) was selected for the chromatographic separation of the components, adjusting the column temperature to 30 °C (LC Ni-II/ADC oven).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Becerro de Bengoa, Phd, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid (Podología), Madrid, Madrid, Spain

REFERENCES:
- [Background] Plusje LG. Pincer nails: a new surgical treatment. Dermatol Surg. 2001 Jan;27(1):41-3. PMID 11231241
- [Background] Baran R, Haneke E, Richert B. Pincer nails: definition and surgical treatment. Dermatol Surg. 2001 Mar;27(3):261-6. PMID 11277894
- [Result] Gao W, Legido-Quigley C. Fast and sensitive high performance liquid chromatography analysis of cosmetic creams for hydroquinone, phenol and six preservatives. J Chromatogr A. 2011 Jul 15;1218(28):4307-11. doi: 10.1016/j.chroma.2011.04.064. Epub 2011 May 6. PMID 21621212